CLINICAL TRIAL: NCT04904640
Title: Evaluation of the Reconstruction of Biomechanical Parameters Provided by Three Different Hip Stem Designs in Developmental Hip Dysplasia Using a 3D CT-based Software for Surgical Planning
Brief Title: Biomechanical Reconstruction of Three Different Hip Stem Designs in Hip Dysplasia Using a 3D CT-based Planning Software
Acronym: CTdevice
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 29/2021/Oss/IOR
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-02

CONDITIONS: Dysplasia; Hip
Keywords: Hip arthroplasty; Hip stem; Pre-operative planning; Combined anteversion; Offset; Developmental dysplasia of the hip
MeSH Terms: conditions — Hip Dislocation; Developmental Dysplasia of the Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CLS stem: CLS Zimmer stem implantation (single wedge, tapered stem) using the 3D CT based software for surgical pre-operative planning
  Interventions: Device: Hip stem
- Wagner cone stem: Wagner cone Zimmer stem implantation (conical tapered stem) using the 3D CT based software for surgical pre-operative planning
  Interventions: Device: Hip stem
- Aptafix stem: Aptafix Ortho stem implantation (anatomical stem) using the 3D CT based software for surgical pre-operative planning
  Interventions: Device: Hip stem

INTERVENTIONS:
Device: Hip stem — In every hip (with appropriate CT scan), 3 different stem designs will be positioned using a 3D Ct based software for surgical pre-operative planning.

SUMMARY:
A random population of 200 CT scans of pelvis and thigh in an adult population affected by hip dysplasia will be selected. The aim of this study is to evaluate the biomechanical reconstruction of the hip anatomy provided by three different hip stem designs in dysplastic cases, using a 3D CT based software for pre-operative planning.

DETAILED DESCRIPTION:
Pre-operative planning in hip arthroplasty with dedicated software is a useful guide to provide a better reconstruction of the biomechanical parameters of the replaced hip and to optimize the choice of component, improving the geometric understanding of the hip anatomy and the interaction between the native morphological structure and the prosthetic component.

The use of a 3D CT-based software for pre-operative planning may provide a better knowledge of the hip anatomy, simulating the biomechanical parameters more closely than a 2D X-ray-based software. In addition, it is the only way to anticipate the correct interaction between the prosthetic components, or the combined anteversion, a key factor in preventing implant instability.

Severe hip deformities, like developmental hip dysplasia, may not be adequately reconstructed by every implant and 3D pre-operative CT may increase the three-dimensional anatomical knowledge of the hip, improving the choice of the correct implant and possibly reducing the possible consequences of intra and post-operative complications.

Therefore, the purpose of this study is to pre-operatively plan, in a random series of 200 native pelvis and thigh CT scans performed in patients with hip dysplasia, 3 different types of hip stem designs using the 3D Hip-Op software, with the aim of analyzing, on the CT simulations, the percentage of adequate reconstruction of the optimal biomechanical parameters (combined anteversion between 25°-50°, global offset not inferior to 12% of the native offset, leg lengthening not superior to 3 cm, sagittal and coronal tilt not superior to +/-5°, canal filling not inferior to 80%). The percentage of every stem design providing the optimal reconstruction in dysplastic hips (all the 5 parameters matched) will be assessed. The single parameters, especially the combined anteversion, the offset restoration and the leg lengthening, will be assessed for every simulation.

ELIGIBILITY:
Inclusion Criteria:

* definition of developmental hip dysplasia according to Wiberg (center edge angle <20°)
* pre-operative CT scan extended from the fourth lumbar vertebra to the tibial plateaus

Exclusion Criteria:

* other types of hip pathologies
* inadequate Ct scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A random population of 200 CT scans (from the fourth lumbar vertebra to the tibial plateaus) involving adult patients with developmental hip dysplasia.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Traina, Professor, Study Director — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- Chirurgia Protesica e dei Reimpianti di Anca e Ginocchio, IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taniguchi N, Jinno T, Koga D, Hagino T, Okawa A, Haro H. Cementless Hip Stem Anteversion in the Dysplastic Hip: A Comparison of Tapered Wedge vs Metaphyseal Filling. J Arthroplasty. 2017 May;32(5):1547-1552. doi: 10.1016/j.arth.2016.12.020. Epub 2016 Dec 22. PMID 28110848
- [Background] Argenson JN, Ryembault E, Flecher X, Brassart N, Parratte S, Aubaniac JM. Three-dimensional anatomy of the hip in osteoarthritis after developmental dysplasia. J Bone Joint Surg Br. 2005 Sep;87(9):1192-6. doi: 10.1302/0301-620X.87B9.15928. PMID 16129740
- [Background] Sugano N, Takao M, Sakai T, Nishii T, Miki H. Does CT-based navigation improve the long-term survival in ceramic-on-ceramic THA? Clin Orthop Relat Res. 2012 Nov;470(11):3054-9. doi: 10.1007/s11999-012-2378-4. PMID 22569720
- [Background] Castagnini F, Valente G, Crimi G, Taddei F, Bordini B, Stea S, Toni A. Component positioning and ceramic damage in cementless ceramic-on-ceramic total hip arthroplasty. J Orthop Sci. 2019 Jul;24(4):643-651. doi: 10.1016/j.jos.2018.12.011. Epub 2019 Jan 4. PMID 30612885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Random selection of pre-operative Ct including native dysplastic hips
Pre-assignment Details: All the 150 patients enrolled in the study underwent a preoperative planning with a particular software, and each hip (200) was studied with three different stem design, so each of them results enrolled in each arm group which represents a different kind of hip stem.
Units Other Than Participants: Hips
Groups:
- Simulated Hips: Hip stem: In every hip (with appropriate CT scan), 3 different stem designs will be positioned using a 3D Ct based software for surgical pre-operative planning.The Three stems are: CLS Zimmer, Wagner Cone Zimmer, Aptafix Adler
Period: Overall Study
Arm/Group | Simulated Hips
Started | 150; 200 Hips
Completed | 150; 200 Hips
Not Completed | 0; 0 Hips

BASELINE CHARACTERISTICS:
Population: All the 150 patients enrolled in the study underwent a preoperative planning with a particular software, and every eligible dysplastic hip (200) was studied with three different stem design
Units Other Than Participants: Hips
Groups:
- Simulated Hips: Hip stem: In every hip (with appropriate CT scan), 3 different stem designs will be positioned using a 3D Ct based software for surgical pre-operative planning. The three stems are: CLS Zimmer (single wedge, tapered stem), Wagner Cone Zimmer (tapered stem), Aptafix Adler (anatomical stem)
Arm/Group | Simulated Hips
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 150
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: hips] — Population: All the 150 patients enrolled in the study underwent a preoperative planning with a particular software, and each hip (200) was studied with three different stem design, so each of them results enrolled in each arm group which represents a different kind of hip stem.
  hips
    Italy | 150
height [Mean (Standard Deviation); unit: centimeters] | 159.8 (18.3)
weight [Mean (Standard Deviation); unit: kg] | 66.1 (15.3)
BMI [Mean (Standard Deviation); unit: kg/m²] | 25.8 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Correct Reconstruction CLS
Description: Percentage of hips correctly reconstructed using CLS stem: the correctly reconstructed hip should have combined anteversion between 25° and 50°, global offset not inferior to 12% of the native offset, leg lengthening not superior to 3 cm, sagittal and coronal tilt not superior to +/-5°, canal filling not inferior to 80% (all the 5 parameters should be present at the same time). Minimum-maximum values (as percentage %): 0-100. 100 is the best result, 0 the worst
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | CLS Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 138

2. Primary Outcome: Correct Reconstruction Wagner Cone
Description: as for outcome 1
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Wagner Cone Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 174

3. Primary Outcome: Correct Reconstruction Aptafix
Description: as for outcome 1
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Aptafix Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 88

4. Secondary Outcome: Combined Anteversion CLS
Description: Percentage of hips with adequate combined anteversion according to Dorr (25-50°) and Widmer (<37°) using CLS stems. Minimum-maximum values (as percentage %): 0-100. 100 is the best result, 0 is the worst
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | CLS Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 153

5. Secondary Outcome: Combined Anteversion Wagner Cone
Description: as for outcome 4
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Wagner Cone Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 197

6. Secondary Outcome: Combined Anteversion Aptafix
Description: as for outcome 4
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Aptafix Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 121

7. Secondary Outcome: Offset CLS
Description: Percentage of hips with acetabular+femoral offset not inferior to 12% of the native value using CLS stems. Minimum-maximum values (as percentage %): 0-100. 100 is the best result, 0 is the worst
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | CLS Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 192

8. Secondary Outcome: Offset Wagner Cone
Description: as for outcome 7
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Wagner Cone Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 186

9. Secondary Outcome: Offset Aptafix
Description: as for outcome 7
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Aptafix Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 164

10. Secondary Outcome: Leg Lengthening CLS
Description: Percentage of hips with leg lengthening not superior to 3 cm using CLS stems. Minimum-maximum values (as percentages %): 0-100. 100 is the best result, 0 is the worst
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | CLS Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 188

11. Secondary Outcome: Leg Lengthening Wagner Cone
Description: as for outcome 10
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Wagner Cone Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 194

12. Secondary Outcome: Leg Lengthening Aptafix
Description: as for outcome 10
Time Frame: Day 0
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Aptafix Stem
Number analyzed (Participants) | 150
Number analyzed (Hips) | 200
Hips | 183

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not assessed
Description: No adverse events were reported, results of the article are based on a prosthetic implants planning software performed on CT scan images.
Arm/Group | CLS Stem | Wagner Cone Stem | Aptafix Stem
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT04904640/Prot_SAP_000.pdf